CLINICAL TRIAL: NCT04733131
Title: Long-term Outcomes After Conversion to a Belatacept-based Immunosuppression in Kidney Transplant
Brief Title: Long-term Outcomes After Conversion to Belatacept
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Paris Translational Research Center for Organ Transplantation (Other)
Responsible Party: Sponsor
Other Study IDs: switch_bela2021
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Kidney Transplant Failure and Rejection; Immunosuppression; Graft Loss; Drug Effect Prolonged
Keywords: belatacept; multicenter study; Long term outcomes
MeSH Terms: conditions — Rejection, Psychology | interventions — Abatacept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- converted to a belatacept based immunosuppression: Belatacept: infusion on Days 1, 15, 29, 43, 57 then every 28 days. All patients received a background maintenance immunosuppressive regimen of mycophenolate mofetil or mycophenolic acid, with adjunctive corticosteroids, according to their immunosuppressive regimen at the time of enrollment.
  Interventions: Drug: Conversion to a belatacept regimen

INTERVENTIONS:
Drug: Conversion to a belatacept regimen — belatacept intravenous on Days 1, 15, 29, 43, 57 then every 28 days.
  Other Names: Nulojix

SUMMARY:
belatacept is a selective T-cell co-stimulation blocker that was approved by Food and Drug Administration (FDA) in 2011 for the prophylaxis of graft rejection in adult kidney transplant recipients. This treatment is indicated as an alternative to Calcineurin Inhibitors (CNIs) for prophylaxis of graft rejection in de novo renal transplant recipients. Long term efficacy and safety outcomes of a kidney transplant population converted to a belatacept regimen after transplant have not been yet reported.

DETAILED DESCRIPTION:
belatacept is a selective T-cell co-stimulation blocker that was approved by Food and Drug Administration (FDA) in 2011 for the prophylaxis of graft rejection in adult kidney transplant recipients. This treatment is indicated as an alternative to Calcineurin Inhibitors (CNIs) for prophylaxis of graft rejection in de novo renal transplant recipients. Major studies evaluating belatacept showed that de novo kidney transplant patients treated with belatacept presented an improved renal function with a higher average estimated glomerular filtration rate (eGFR) compared to ciclosporin (CsA) regimen in patients. Conversion to belatacept after transplant seems to be safe even in highly sensitized patients. However, long term efficacy and safety outcomes of a kidney transplant population converted to a belatacept regimen after transplant and compared to a matched control group under a CNIs regimen have not been yet reported.

A multicenter cohort of kidney transplant patients, will be use to match patients converted to a belatacept immunosuppressive regimen to a control group under CNIs immunosuppressive regimen.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female, over 18 years of age
* Recipient of kidney allograft from a living donor or a deceased donor

Exclusion Criteria:

* Graft loss during the first three months post-transplant
* Epstein-Barr virus Seronegative in the belatacept group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients converted to a belatacept regimen after kidney transplant
Sampling Method: Non-Probability Sample
Enrollment: 324 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2021-06 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Allograft survival after conversion to belatacept | 5 years
  Graft loss is defined as either functional loss or physical loss (nephrectomy). Functional loss is defined as an eGFR< 15 ml/min/1.73m2 or consecutive days of dialysis. For patients who died with a functioning graft, graft survival will be censored at the time of death as a survived or functional graft.
Patient survival after conversion to belatacept | 5 years
  Patient survival after conversion to a belatacept regimen

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Loupy, MD, PhD, Principal Investigator — Paris Translational Research Center for Organ Transplantation

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Divard G, Aubert O, Debiais-Deschamp C, Raynaud M, Goutaudier V, Sablik M, Sayeg C, Legendre C, Obert J, Anglicheau D, Lefaucheur C, Loupy A. Long-Term Outcomes after Conversion to a Belatacept-Based Immunosuppression in Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2024 May 1;19(5):628-637. doi: 10.2215/CJN.0000000000000411. Epub 2024 Feb 22. PMID 38265815